CLINICAL TRIAL: NCT05908734
Title: A Phase 1/2 Study Evaluating the Safety and Efficacy of Amivantamab and Cetrelimab Combination Therapy in Metastatic Non-small Cell Lung Cancer
Brief Title: A Study of Combination Therapy With Amivantamab and Cetrelimab in Participants With Metastatic Non-small Cell Lung Cancer
Acronym: PolyDamas
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109323; 61186372PANSC2002 (Other: Janssen Research & Development, LLC); 2022-501452-29-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-06-06; First posted 2023-06-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Combination Dose Selection) (Experimental): Participants will receive amivantamab low dose or high dose intravenous (IV) infusion based on body weight from Cycle 1 Day 1, Day 2, and subsequently Day 8, Day 15, and Day 22 and then every 2 weeks from Cycle 2 in combination with cetrelimab IV infusion from Cycle 1 Day 2 (after the Day 2 infusion of amivantamab). Cetrelimab treatment duration will be limited to a maximum of 24 months. Doses will be escalated or de-escalated based on the dose limiting toxicities (DLTs) and the recommended Phase 2 combination dose (RP2CD) will be determined by the study evaluation team (SET). Participants who continue to benefit from study treatment(s), as determined by their investigator, may continue to receive access to study treatment(s) within the study by transferring to a long term extension (LTE) phase.
  Interventions: Drug: Cetrelimab; Drug: Amivantamab
- Phase 2 (Dose Expansion) (Experimental): Participants will receive amivantamab in combination with cetrelimab in Cohorts A and B at the RP2CD determined by the SET in Phase 1. Participants will continue study treatment until disease progression, unacceptable toxicity, or until another criterion for discontinuation of study treatment is met. Cetrelimab treatment duration will be limited to a maximum of 24 months. Participants who continue to benefit from study treatment(s), as determined by their investigator, may continue to receive access to study treatment(s) within the study by transferring to an LTE phase.
  Interventions: Drug: Cetrelimab; Drug: Amivantamab

INTERVENTIONS:
Drug: Cetrelimab — Cetrelimab will be administered as IV infusion.
  Other Names: JNJ-63723283
Drug: Amivantamab — Amivantamab will be administered as IV infusion.
  Other Names: JNJ-61186372

SUMMARY:
The purpose of this study is to identify the recommended Phase 2 (combination) dose (RP2CD) of the amivantamab and cetrelimab combination therapy in participants with non-small cell lung cancer (NSCLC) in Phase 1 (combination dose selection); and to evaluate the antitumor effect of the combination at the selected RP2CD in participants with NSCLC characterized on the basis of epidermal growth factor receptor (EGFR) and Programmed-cell death Ligand (PD-L)1 status, in the Phase 2 (expansion).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically or cytologically confirmed non-small cell lung cancer (NSCLC) (any histology), and must have metastatic NSCLC at the time of enrollment: Phase 1 (Combination Dose Selection) Cohort; Metastatic NSCLC progressed on or after standard of care systemic anti-cancer therapy and participant is declining other systemic treatment options, if any;1. Participants without known mutations must have had disease progression on, or have intolerance to, prior platinum-based chemotherapy and PD-(L)1-targeted immunotherapy given concurrently or sequentially, OR 2. Participants with NSCLC characterized by known driver mutations must have had disease progression on, or have intolerance to, appropriate targeted therapies as per local standard of care. Participants may have received prior therapy with amivantamab as long as discontinuation was not due to toxicity. Participants with EGFR mutation must not have had an anti-PD-1/PD-L1 therapy, Phase 2 Expansion Cohorts; Cohort A: Participant's tumor must have an EGFR exon19del or L858R mutation, as determined by local molecular testing, Cohort B: Participants must have tumors lacking known primary driver mutations and must have PD-L1 expression of greater than or equal to (>=)50 percentage (%), per local testing, and are treatment-naïve in the metastatic setting
* Participant must have at least 1 measurable lesion, according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, that has not been previously irradiated
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Participant has an uncontrolled illness, including but not limited to: a. Uncontrolled diabetes, b. Ongoing or active infection (includes infection requiring treatment with antimicrobial therapy [participants will be required to complete antibiotics 1 week prior to starting study treatment] or diagnosed or suspected viral infection), c. Active bleeding diathesis, d. Impaired oxygenation requiring continuous oxygen supplementation, e. Psychiatric illness or any other circumstances (including social circumstances) that would limit compliance with study requirements
* Medical history of (non-infectious) interstitial lung disease (ILD)/pneumonitis, or has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Has an active autoimmune disease or a documented history of autoimmune disease that requires systemic steroids or immunosuppressive agents
* Participant has received radiotherapy for palliative purposes less than 14 days prior to the first dose of study treatment
* Participant has a. (or has a history of) leptomeningeal disease (carcinomatous meningitis), b. spinal cord compression not definitively treated with surgery or radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of Participants with Adverse events (AEs) by Severity | Up to 2 years 3 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the intervention. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Phase 1: Number of Participants with Dose Limiting Toxicities (DLTs) | Up to Cycle 1 (Day 1 through Day 28)
  The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, hematological toxicity, pulmonary toxicity, liver enzyme elevation, treatment delay greater than (>) 28 days due to unresolved toxicity, or immune-related toxicity requiring the use of therapies in excess of corticosteroids.
Phase 2: Objective Response Rate | Up to 2 years 3 months
  ORR is defined as the percentage of participants who achieve either a confirmed partial response (PR) or complete response (CR), using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as per investigator assessment.

SECONDARY OUTCOMES:
Phase 1 and Phase 2: Number of Participants with AEs by Severity | Up to 2 years 3 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the intervention. Severity will be graded according to the NCI-CTCAE version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Phase 1 and Phase 2: Number of Participants with Abnormalities in Clinical Laboratory Parameters | Up to 2 years 3 months
  Number of participants with abnormalities in clinical laboratory parameters (serum chemistry, hematology, coagulation, serology, and urinalysis) will be reported.
Phase 2 : Duration of Response (DoR) | Up to 2 years 3 months
  DoR is defined as the time from the date of first documented response (PR or CR) until the date of documented progression or death from any case, whichever comes first, for participants who have PR or CR. If a participant does not progress following a response, then his/her duration of response will be censored at the date of last evaluable disease assessment. Participants who started a subsequent anticancer therapy in the absence of progression will be censored at the last disease assessment before or on the start of subsequent therapy.
Phase 2: Disease Control Rate (DCR) | Up to 2 years 3 months
  DCR is defined as the percentage of participants who achieve a PR, CR, or stable disease using RECIST version 1.1 by investigator review.
Phase 2: Progression Free Survival (PFS) | Up to 2 years 3 months
  PFS is defined as the time from first dose date until the date of disease progression or death, whichever comes first, based on investigator assessment using RECIST version 1.1. Participants who have not progressed or have not died at the time of analysis will be censored at the time of their last evaluable RECIST v1.1 assessment.
Phase 2: Overall Survival (OS) | Up to 2 years 3 months
  OS is defined as the time from the date of administration of the first study treatment until the date of death due to any cause. Any participant not known to have died at the time of analysis will be censored based on the last recorded date on which the participant was known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (44):
- United States (7):
  - City of Hope, Duarte, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Oncology and Hematology Care Clinic Westside, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Brazil (8):
  - Fundacao Pio XII, Barretos
  - Cetus Oncologia, Belo Horizonte
  - PERSONAL Oncologia de Precisao e Personalizada, Belo Horizonte
  - CIONC Centro Integrado de Oncologia de Curitiba, Curitiba
  - Hospital do Cancer de Londrina, Londrina
  - Hospital Nossa Senhora da Conceicao S A, Porto Alegre
  - Hospital Santa Izabel Santa Casa de Misericordia da Bahia, Salvador
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
- Italy (4):
  - European Institute of Oncology, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Aou San Luigi Gonzaga, Orbassano
  - Centro Ricerche Cliniche di Verona S r l, Verona
- Malaysia (2):
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
- Poland (3):
  - INSTYTUT GENETYKI I IMMUNOLOGII GENIM Sp z o o, Lublin
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii im. Eugenii i Janusza Zeylandow, Poznan
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. Quiron Dexeus, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Virgen Macarena, Seville
  - Instituto Valenciano de Oncologia, Valencia
- Turkey (Türkiye) (8):
  - Adana City Hospital, Adana
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Ankara Bilkent City Hospital, Çankaya
  - Bakirkoy Sadi Konuk Training and Research Hospital, Istanbul
  - Goztepe Prof Dr Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Medicana International Izmir, Izmir
  - Sakarya University Training and Research Hospital, Sakarya
- United Kingdom (3):
  - Imperial College London and Imperial College Healthcare NHS Trust, London
  - Freeman Hospital, Newcastle
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency